CLINICAL TRIAL: NCT06721715
Title: Textbook Outcomes After Oesophagectomy in a Regional Australian Hospital: a Retrospective Observational Cohort Study
Brief Title: Textbook Outcomes After Oesophagectomy in Regional Australia
Status: Not yet recruiting | Type: Observational
Sponsor: Launceston General Hospital (Other)
Responsible Party: Principal Investigator, Renishka Sellayah, General Surgery Fellow, Launceston General Hospital
Other Study IDs: 2024/STE03324
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Oesophageal Cancer Nos
Keywords: oesophagectomy; oesophageal cancer; regional surgery
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Textbook outcome: Patients that achieve a textbook outcome after oesophagectomy
- No textbook outcome: Patients who do not achieve a textbook outcome after oesophagectomy

SUMMARY:
The goal of this observational cohort study is to assess textbook outcomes after oesophagectomy in a regional Australian hospital. This is a composite quality measure that include 9 parameters related to cancer care. Researchers will compares the textbook outcome rate in this regional hospital and compare it to textbook outcomes rates from other Australian hospitals, as well as hospitals overseas. Participants will not be actively involved in this study, as all data will be collected from medical records only.

DETAILED DESCRIPTION:
Rationale Textbook outcomes is a composite tool to assess the quality of cancer care within an institution by evaluating several perioperative and postoperative factors. Most studies assessing textbook outcomes after oesophagectomy have been conducted in high-volume centres, achieving rates of up to 50%. To the best of our knowledge this is the first study to assess textbook outcomes after oesophagectomy in a regional Australian hospital, providing a unique insight into the performance of this procedure in a country that has not widely adopted centralisation of cases.

Aims/objectives To calculate textbook outcomes rates in a regional hospital in Australia and compare to higher volume Australian and international institutions.

Methods Retrospective identification of patients from MBS codes related to oesphagectomy, and collection of data retrospectively from the medical record only. All patients undergoing oesophagectomy from January 2014 to December 2023 will be included. There are no exclusion criteria.

Data collection Baseline patient characteristics, tumour-specific factors, textbook outcome parameters, treatment details including postoperative complications, and follow up data on survival will be collected

Statistical analysis Statistical analysis will be performed in consultation with a biostatistician. The number and proportion of patients who meet each parameter of the textbook outcome will be calculated for each year and compared. Patient characteristics (age, gender, BMI and ASA grade), tumour factors (histology, AJCC clinical T and N stage), and treatment aspects (neoadjuvant therapy and surgical approach) will be assessed for association with textbook outcomes using the Chi squared test with significance considered less than 0.05. A Kaplan-Meier survival curve will be used to investigate overall survival of patients with and without a textbook outcome.

ELIGIBILITY:
Inclusion Criteria:

* all patients who underwent oesophagectomy between January 2014 and December 2023

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent oesophagectomy at a single regional hospital in Tasmania, Australia between January 2014 and December 2023 will be included in this study,
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Textbook outcome | from date of surgery to end of study (December 2024) for a timeframe up to 10 years
  Patients who achieve a textbook outcome. This is defined when all 9 following criteria are met: R0 resection, retrieval of 15 or more lymph nodes, no intraoperative complications, no post-operative complications Clavien-Dindo grade III or higher, no readmission to the ICU, no hospital stay longer than 21 days, no mortality within 90 days, no readmission related to the procedure within 30 days of admission, and no reintervention related to the surgical procedure (operative, endoscopic or radiologic).

CONTACTS AND LOCATIONS:
Locations (1):
- Launceston General Hospital, Launceston, Tasmania, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalff MC, Vesseur I, Eshuis WJ, Heineman DJ, Daams F, van der Peet DL, van Berge Henegouwen MI, Gisbertz SS. The Association of Textbook Outcome and Long-Term Survival After Esophagectomy for Esophageal Cancer. Ann Thorac Surg. 2021 Oct;112(4):1134-1141. doi: 10.1016/j.athoracsur.2020.09.035. Epub 2020 Nov 19. PMID 33221197
- [Background] Kay B, Healy TE. Propofol ('Diprivan') for outpatient cystoscopy. Efficacy and recovery compared with althesin and methohexitone. Postgrad Med J. 1985;61 Suppl 3:108-14. PMID 3877277
- [Background] Kalff MC, van Berge Henegouwen MI, Gisbertz SS. Textbook outcome for esophageal cancer surgery: an international consensus-based update of a quality measure. Dis Esophagus. 2021 Jul 12;34(7):doab011. doi: 10.1093/dote/doab011. PMID 33744921
- [Background] Ball ED, Keefe KA, Colby E. Expression of antigens associated with small cell carcinoma of the lung on hematopoietic progenitor cells. Cancer Res. 1987 Dec 15;47(24 Pt 1):6556-9. PMID 2824035
- [Background] van der Werf LR, Wijnhoven BPL, Fransen LFC, van Sandick JW, Nieuwenhuijzen GAP, Busweiler LAD, van Hillegersberg R, Wouters MWJM, Luyer MDP, van Berge Henegouwen MI. A National Cohort Study Evaluating the Association Between Short-term Outcomes and Long-term Survival After Esophageal and Gastric Cancer Surgery. Ann Surg. 2019 Nov;270(5):868-876. doi: 10.1097/SLA.0000000000003520. PMID 31634182